CLINICAL TRIAL: NCT03643211
Title: XELJANZ(REGISTERED) TABLETS 5 MG SPECIAL INVESTIGATION(INVESTIGATION OF LONG-TERM USE IN PATIENTS WITH ULCERATIVE COLITIS)
Brief Title: Xeljanz Special Investigation for Long-term Use in UC Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921248
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis
Keywords: Xeljanz; Ulcerative colitis; UC; Long-term
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Secondary data collection study: safety and effectiveness of Xeljanz in UC patients under Japanese medical practice

DETAILED DESCRIPTION:
This investigation aims to examine the safety and effectiveness of Xeljanz in post-marketing clinical settings when it is administered chronically to patients with ulcerative colitis, based on the approval conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ulcerative colitis treated with XELJANZ
* Patients naive to XELJANZ in the treatment of ulcerative colitis

Exclusion Criteria:

- None

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: UC patients who were confirmed to have received Xeljanz after the approval date of dosage and administration of Xeljanz for UC patients
Sampling Method: Probability Sample
Enrollment: 2016 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Local Country Office, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Matsuoka K, Motoya S, Shinzaki S, Mikami Y, Adachi C, Arai S, Endo Y, Sato K, Yuasa H, Mizuno Y, Hisamatsu T. Post-marketing Surveillance of Tofacitinib in Patients With Ulcerative Colitis in Japan: A Post Hoc Analysis of Safety and Effectiveness by Prior Biologic Status. Crohns Colitis 360. 2025 Nov 22;7(4):otaf065. doi: 10.1093/crocol/otaf065. eCollection 2025 Oct. PMID 41425505
- [Derived] Matsuoka K, Motoya S, Yamamoto T, Matsuura M, Fujii T, Shinzaki S, Mikami Y, Arai S, Oshima J, Endo Y, Yuasa H, Hoshi M, Sato K, Hisamatsu T. Post-marketing surveillance of tofacitinib in patients with ulcerative colitis in Japan: a final report of safety and effectiveness data. J Gastroenterol. 2025 Aug;60(8):979-989. doi: 10.1007/s00535-025-02249-5. Epub 2025 Apr 21. PMID 40259041
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921248

RESULTS

PARTICIPANT FLOW:
Groups:
- XELJANZ Tablets 5 mg (Tofacitinib Citrate): Participants who received XELJANZ as indicated in the approved local product document were observed for a period of 60 weeks. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | XELJANZ Tablets 5 mg (Tofacitinib Citrate)
Started | 2016
Completed | 1995
Not Completed | 21
Not completed — Contract violation/deficiency | 12
Not completed — Invalid registration | 3
Not completed — No treatment information | 2
Not completed — No adverse event information - No revisit | 4

BASELINE CHARACTERISTICS:
Population: A total of 2016 participants were enrolled in this study. Of the 2016 participants from whom CRFs were collected, 21 participants were excluded from the safety analysis set due to the following reasons: contract violation/deficiency (12 participants), invalid registration (3 participants), no treatment information (2 participants), and no adverse event information - no revisit (4 participants).
Arm/Group | XELJANZ Tablets 5 mg (Tofacitinib Citrate)
Number analyzed (Participants) | 1995
Age, Customized [Number; unit: Participants]
  <15 years | 12
  ≥15 and <65 years | 1770
  ≥65 years | 213
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 782
  Male | 1208
  Unknown | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to XELJANZ in a participant who received XELJANZ. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to XELJANZ was assessed by the physician.
Time Frame: 60 weeks
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received XELJANZ at least once. Participants with contract violation/deficiency, invalid registration, no treatment information, and no adverse event information - no revisit were excluded.
Measure: Number; unit: Participants
Arm/Group | XELJANZ Tablets 5 mg (Tofacitinib Citrate)
Number analyzed (Participants) | 1995
Participants
  ADR | 466
  Serious ADR | 46

ADVERSE EVENTS:
Time Frame: 60 weeks
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | XELJANZ Tablets 5 mg (Tofacitinib Citrate)
All-Cause Mortality (participants affected / at risk) | 1/1995
Serious Adverse Events (participants affected / at risk) | 103/1995
Other Adverse Events (participants affected / at risk) | 586/1995
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XELJANZ Tablets 5 mg (Tofacitinib Citrate) (N=1995)
Anaemia (Blood and lymphatic system disorders) | 3
Myelosuppression (Blood and lymphatic system disorders) | 1
Retinal detachment (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Anal fistula (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 30
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Rectal perforation (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Drug ineffective (General disorders) | 2
Dysplasia (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 8
Therapeutic response decreased (General disorders) | 6
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1
Abscess intestinal (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Atypical mycobacterial infection (Infections and infestations) | 2
Bone tuberculosis (Infections and infestations) | 1
Clostridium colitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 1
Cytomegalovirus enterocolitis (Infections and infestations) | 2
Cytomegalovirus infection (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 1
Eczema herpeticum (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 4
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Carcinoembryonic antigen increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Encephalopathy (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Aortic dissection (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XELJANZ Tablets 5 mg (Tofacitinib Citrate) (N=1995)
Anaemia (Blood and lymphatic system disorders) | 26
Anaemia macrocytic (Blood and lymphatic system disorders) | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 11
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Neutrophilia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Palpitations (Cardiac disorders) | 2
Type IIa hyperlipidaemia (Congenital, familial and genetic disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Meniere's disease (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain lower (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 3
Anal erosion (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Appendiceal mucocoele (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 35
Colon dysplasia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 2
Gastric polyps (Gastrointestinal disorders) | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival swelling (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 3
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Leukoplakia oral (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mouth swelling (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Pancreatitis acute (Gastrointestinal disorders) | 1
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 5
Chest pain (General disorders) | 2
Chills (General disorders) | 1
Drug ineffective (General disorders) | 5
Dysplasia (General disorders) | 1
Generalised oedema (General disorders) | 1
Malaise (General disorders) | 18
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 2
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 27
Therapeutic product effect incomplete (General disorders) | 1
Therapeutic response decreased (General disorders) | 10
Cholestasis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 28
Hepatic steatosis (Hepatobiliary disorders) | 3
Liver disorder (Hepatobiliary disorders) | 15
Anal abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 2
Clostridium difficile infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Cytomegalovirus infection (Infections and infestations) | 3
Device related infection (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 6
Enterocolitis viral (Infections and infestations) | 2
Folliculitis (Infections and infestations) | 2
Fungal skin infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis bacterial (Infections and infestations) | 1
Gastroenteritis norovirus (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Genital herpes simplex (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 90
Infectious mononucleosis (Infections and infestations) | 1
Influenza (Infections and infestations) | 10
Nasopharyngitis (Infections and infestations) | 24
Norovirus infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 9
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 6
Pneumonia bacterial (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Rubella (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Tinea cruris (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Varicella (Infections and infestations) | 2
Rib fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 5
Blood albumin decreased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 3
Blood beta-D-glucan increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 4
Blood creatine phosphokinase increased (Investigations) | 22
Blood creatinine increased (Investigations) | 6
Blood glucose abnormal (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Blood potassium increased (Investigations) | 2
Blood pressure increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 3
Blood urea increased (Investigations) | 1
Clostridium test positive (Investigations) | 1
Cortisol decreased (Investigations) | 1
C-reactive protein increased (Investigations) | 5
Gamma-glutamyltransferase increased (Investigations) | 3
Glomerular filtration rate decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 4
Hepatic enzyme increased (Investigations) | 2
KL-6 increased (Investigations) | 1
Lipids abnormal (Investigations) | 5
Low density lipoprotein increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 12
Macroenzyme creatine kinase (Investigations) | 1
Mean cell volume decreased (Investigations) | 1
Mean cell volume increased (Investigations) | 1
Monocyte count increased (Investigations) | 2
Monocyte percentage increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 8
Neutrophil count increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 8
White blood cell count increased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 5
Dyslipidaemia (Metabolism and nutrition disorders) | 20
Hypercholesterolaemia (Metabolism and nutrition disorders) | 20
Hypercreatininaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 30
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Zinc deficiency (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chondritis (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
SAPHO syndrome (Musculoskeletal and connective tissue disorders) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 25
Hypoaesthesia (Nervous system disorders) | 2
Loss of consciousness (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Taste disorder (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Abortion of ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Adjustment disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Dysphoria (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Calculus urinary (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 3
Ureterolithiasis (Renal and urinary disorders) | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 10
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 4
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 16
Urticaria (Skin and subcutaneous tissue disorders) | 8
Tooth extraction (Surgical and medical procedures) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 8
Peripheral coldness (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 2
Venous thrombosis limb (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT03643211/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT03643211/SAP_001.pdf